CLINICAL TRIAL: NCT04125407
Title: The Effect of Sensorimotor Insoles on Gait Parameters in Adults With Flexible Flatfoot: A Randomised Control Trial
Brief Title: The Effect of Sensorimotor Insoles on Gait Parameters in Adults With Flexible Flatfoot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Zdenek Svoboda, Assistant Professor, Palacky University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UPOL_FTK_2019_007
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Flexible Flatfoot
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Experimental group will receive one customized pair of sensorimotor foot orthoses (insoles).
  Intervention: Other: Sensorimotor foot orthoses with any other supplementary treatment.
  Interventions: Other: Sensorimotor foot orthoses
- Control (No Intervention): Control group will receive neither orthotic nor other supplementary intervention.

INTERVENTIONS:
Other: Sensorimotor foot orthoses — The interventional group will receive one customized pair of sensorimotor insoles and will be instructed for their using on a daily bases for the period of 3 months. The duration of using the insoles was established as 1 hour at the day after receiving the insoles. After that, the insoles' tolerance will be assessed based on the email correspondence and further adjustments of insole will be consulted with manufacturer if necessary. Recommended progression in time of using the insoles was established as +1 hour per each day (if possible) with no maximal limit. After 3 weeks, control examination will take place for the control of subjective effect of insoles. Consulting will be offered to the participants through the duration of research. Participants will not undergo any other supplementary treatment (physiotherapy, …) focusing on the flatfoot deformity.
  Arms: Interventional

SUMMARY:
The flatfoot is one of the most common diagnosis in foot. The main goals of its orthotic intervention in adult population are the control of the rearfoot and midfoot movement, the affection of the forefoot position and the minimalization of painful deformities. However, only low-level evidence exists proving the positive effect of orthotic insoles in these patients. The concept of sensorimotor insoles describes besides the simple mechanical correction also the targeted modulation of activity of muscles participated on the correct foot function. The aim of the project is to assess the influence of customized sensorimotor insoles on the lower limbs' kinematics and the activity of lower limbs' muscles in people with diagnosed flexible flatfoot.

The study is designed as a crossover interventional study with experimental and control group (allocation ratio 1:1). Participants' lower limbs' kinematics and muscles activity will be assessed on the baseline measurement, immediately after and 3 months after the intervention with sensorimotor insoles in the experimental group. Also, the subjective perceived effect of intervention will be assessed through the research. After a washout period, experimental and control group will swap their roles and another period of 3 months will follow. Same parameters will be assessed both at the beginning and in the end of each period.

ELIGIBILITY:
Inclusion Criteria:

* ability to stand and walk without aid or support
* flat foot deformity confirmed by the Foot Posture Index (FPI-6) score >5 and/or the normalised navicular height truncated <0.21

Exclusion Criteria:

* congenital and/or acquired neuromuscular or orthopaedic impairments that severely limit mobility and/or balance
* any acute pain while standing and/or walking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Foot kinematics - difference in foot eversion relative to shank during the stance phase of the gait cycle | 3 months
  The two-way analysis of variance of the degree of the first peak of foot eversion measured by the optoelectronic system Vicon Vantage (Vicon Motion Systems Ltd., Oxford, Great Britain), where the factors are the "group" (intervention, control) and "time" (baseline, after 3 months).
Foot kinematics - difference in foot external rotation relative to shank during the stance phase of the gait cycle | 3 months
  The two-way analysis of variance of the degree of the first peak of foot external rotation measured by the optoelectronic system Vicon Vantage (Vicon Motion Systems Ltd., Oxford, Great Britain), where the factors are the "group" (intervention, control) and "time" (baseline, after 3 months).

SECONDARY OUTCOMES:
Surface electromyography - difference in muscle activity by parameter "mean" during the stance phase of the gait cycle | 3 months
  The two-way analysis of variance of the mean activity of the tibialis anterior, peroneus longus and gastrocnemius medialis muscles measured by the TrignoTM Wireless Systems (Delsys Inc., Natick, MA, USA) and normalised to their peak activity during the stance phase of the gait cycle, where the factors are the "group" (intervention, control) and "time" (baseline, after 3 months).

OTHER OUTCOMES:
Global Rating of Change Scale | 3 months
  Subjective evaluation of overall change in health status on the 11-point scale after 3 month from the baseline, where 0 means "unchanged", -5 means "very much worse" and +5 means "completely recovered".

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Lastovicka, Study Director — Faculty of Physical Culture, Palacky University Olomouc
Locations (1):
- Faculty of Physical Culture, Palacky University Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No